CLINICAL TRIAL: NCT02672735
Title: Influence of a Corrective Exercise Training Program on Measures of Functional Movement Among Active-Duty Firefighters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Kyle T Ebersole, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.389
Record Dates: First submitted 2015-08-27; First posted 2016-02-03 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Functional Movement Quality
Keywords: corrective exercise program; movement efficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corrective Exercise Program (Experimental): Participants in the Corrective Exercise Program (CEP) group (n = 28) will be given a four-week corrective exercise programming intervention.
  Interventions: Other: Corrective Exercise Programming
- Control (No Intervention): The participants in the Control (CON) group (n = 28) will have their four-week corrective exercise programming intervention deferred for 4 weeks, and as such, will serve as the comparative group for the CEP group.

INTERVENTIONS:
Other: Corrective Exercise Programming — Participants will be given a four-week corrective exercise protocol, with four corrective exercise sessions prescribed each week. Participants in the CEP Group will be required to complete a minimum of three of these four training sessions per week throughout the four-week corrective exercise program intervention. All corrective exercise programming will be created through the Fusionetics Human Performance System. This system, along with weekly compliance questionnaires, will also assess the compliance-level among the participants.
  Arms: Corrective Exercise Program

SUMMARY:
The occupation of firefighting is considered to be one of the most dangerous occupations in the United States (U.S.). As such, a high prevalence of musculoskeletal injuries (MSKIs) have been observed among the firefighter population. This high rate of MSKI has created an extremely large financial impact on fire departments across the United States. Therefore, interest in developing methods of identifying those at risk for developing a future MSKI and interventions designed to prevent these MSKIs from happening has grown among both the firefighter population, as well as among researchers and practitioners.

Previous research has demonstrated relationships between MSKI and altered movement patterns. In addition, researchers have started to demonstrate the ability of functional movement assessments to predict future MSKI in various populations, including firefighters. Two of these functional movement assessments include the Functional Movement Screen (FMS) and the Movement Efficiency (ME) Test, which is a component of the Fusionetics Human Performance System. These assessments both quantify the overall functional movement quality of an individual by creating a composite movement score (i.e., Total FMS & Average ME Test scores, respectively).

In addition, various theoretical models of corrective exercise programming have been proposed. These programs are designed to restore optimal neuromuscular control and correct any identified neuromuscular imbalances observed during the movement assessment through the use of simple and easy-to-follow exercises. The Fusionetics Human Performance System utilizes one such model, with the goal of improving the functional movement quality of an individual by correcting the aforementioned neuromuscular deficiencies observed during the ME Test. Based on this framework, these corrective exercise programs theoretically lower the risk of MSKI of the individual as well.

However, there is currently a lack of research in the literature examining the influence of corrective exercise programming on functional movement quality among the active-duty firefighter population. As such, it remains unknown if a corrective exercise intervention is capable of significantly improving functional movement quality among active-duty firefighters. In addition, recent research suggests that various health and fitness measures are associated with functional movement quality. These measures include total body power output, lower extremity muscular strength, and core muscular endurance. As such, an examination of the influence of a corrective exercise intervention on measures of health and fitness among active-duty firefighters is warranted.

ELIGIBILITY:
General Eligibility Criteria:

Participants will be considered eligible for this study if they:

1. are fluent in speaking and writing English;
2. are at least 18 years of age;
3. they are an active-duty firefighter;
4. are cleared by their fire department for full active-duty work; and
5. have been an active-duty firefighter for at least 12 months (i.e., one year).

Inclusion Criteria:

Participants will be included into this study if they:

1. do not suffer from chest pain or dizziness;
2. have not been diagnosed with a heart condition;
3. are not currently pregnant;
4. have not had any serious ankle, knee, hip, back, or shoulder trauma that required medical attention in the past 3 months;
5. have not had surgery on their ankle, knee, hip, back, or shoulder within the past year (12 months); or
6. do not have any current bone, joint, or muscle abnormalities that require medical attention;
7. have not been instructed by a physician or their Health and Safety Officer (HSO) to not participate in this study.

Exclusion Criteria:

1. Participants will be excluded from being placed into Phase 2 (i.e., the intervention portion) of this study if they are already engaged in a structured corrective exercise program. Furthermore, in order to ensure similar baseline functional movement quality between the CEP and CON groups, participants will be excluded from being placed into the intervention portion of this study if their Overall MET score is < 25 or > 75.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in Total Functional Movement Screen (FMS) Score | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  The Functional Movement Screen (FMS) is a seven task movement screen test that will be scored on a 4-point scale (0-3, worst-best), for a total of 21 possible points.
Change in Overall Movement Efficiency (ME) Test Score | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  The Movement Efficiency (ME) Test, which is part of the Fusionetics Human Performance System, uses a 0-100 scale to score the functional movement quality of an individual.
Change in Dynamic Balance Ability | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  The dynamic balance ability of each participant will be assessed by utilizing the Y-Balance Test (YBT).

SECONDARY OUTCOMES:
Change in Range of Motion | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  Passive range of Motion (PROM) for the foot, ankle, knee, hip, shoulder, and trunk will be bilaterally measured with a standard plastic goniometer (a kind of ruler).
Change in Total Body Power Output | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  Total body power output will be examined by performing a countermovement jump (CMJ), which is a field-test commonly utilized by practitioners to examine total body power output.
Change in Lower Extremity Isometric Muscular Strength | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  The isometric lower extremity muscular strength of each participant will be examined utilizing the Jackson Strength Evaluation System.
Change in Core Muscular Endurance | Pre-Intervention (Week 0), Mid-Intervention (Week 3), Post-Intervention (Week 5)
  The overall core muscular endurance of each participant will be examined through the use of a prone plank. Participants will perform a prone plank until volitional fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle T. Ebersole, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Station 5, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton, L., Kiesel, K., & Cook, G. (2004). Mobility screening for the core: Interventions. Athletic Therapy Today, 9(6), 52-57.
- [Background] Butler RJ, Contreras M, Burton LC, Plisky PJ, Goode A, Kiesel K. Modifiable risk factors predict injuries in firefighters during training academies. Work. 2013 Jan 1;46(1):11-7. doi: 10.3233/WOR-121545. PMID 23324700
- [Background] Clark, M.A, & Lucett, S.C. (2011). NASM Essentials of Corrective Exercise Training (1st ed.). Baltimore, MD: Lippincott Williams & Wilkins.
- [Background] Comerford MJ, Mottram SL. Functional stability re-training: principles and strategies for managing mechanical dysfunction. Man Ther. 2001 Feb;6(1):3-14. doi: 10.1054/math.2000.0389. PMID 11243904
- [Background] Comerford MJ, Mottram SL. Movement and stability dysfunction--contemporary developments. Man Ther. 2001 Feb;6(1):15-26. doi: 10.1054/math.2000.0388. PMID 11243905
- [Background] Cook, G. (2003). Athletic Body in Balance. Champaign, IL: Human Kinetics.
- [Background] Cook, G. (2010). Movement: Functional Movement Systems - Screening, Assessment and Corrective Strategies. Santa Cruz, CA: On Target Publications.
- [Background] Cook G, Burton L, Hoogenboom BJ, Voight M. Functional movement screening: the use of fundamental movements as an assessment of function - part 1. Int J Sports Phys Ther. 2014 May;9(3):396-409. PMID 24944860
- [Background] Cook G, Burton L, Hoogenboom BJ, Voight M. Functional movement screening: the use of fundamental movements as an assessment of function-part 2. Int J Sports Phys Ther. 2014 Aug;9(4):549-63. PMID 25133083
- [Background] Duncan MJ, Stanley M. Functional movement is negatively associated with weight status and positively associated with physical activity in british primary school children. J Obes. 2012;2012:697563. doi: 10.1155/2012/697563. Epub 2012 Mar 26. PMID 22545208
- [Background] Duncan MJ, Stanley M, Leddington Wright S. The association between functional movement and overweight and obesity in British primary school children. BMC Sports Sci Med Rehabil. 2013 May 15;5:11. doi: 10.1186/2052-1847-5-11. eCollection 2013. PMID 23675746
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Harman, E., & Garhammer, J. (2008). Administration, scoring, and interpretation of selected tests. In T.R. Baechle, & R.W. Earle (Eds.), Essentials of Strength Training and Conditioning (3rd ed., pp. 250-292). Champaign, IL: Human Kinetics.
- [Background] Hirth, C.J. (2007). Clinical movement analysis to identify muscle imbalances and guide exercise. Athletic Therapy Today, 12(4), 10-14.
- [Background] International Association of Fire Fighters. (2008). The Fire Service Joint Labor Management Wellness-Fitness Initiative, (3rd ed.). Washington, D.C.
- [Background] Kiesel, K, Burton, L., & Cook, G. (2004). Mobility screening for the core. Athletic Therapy Today, 9(5), 38-41.
- [Background] Knapik JJ, Cosio-Lima LM, Reynolds KL, Shumway RS. Efficacy of functional movement screening for predicting injuries in coast guard cadets. J Strength Cond Res. 2015 May;29(5):1157-62. doi: 10.1519/JSC.0000000000000704. PMID 25264669
- [Background] Kritz, M., Cronin, J., & Hume, P. (2009). The bodyweight squat: A movement screen for the squat pattern. Strength and Conditioning Journal, 31(1), 76-85.
- [Background] Kritz, M., Cronin, J., & Hume, P. (2009). Using the body weight forward lunge to screen an athlete's lunge pattern. Strength and Conditioning Journal, 31(6), 15-24.
- [Background] Kurlick G.M. (2012). Stop, drop, and roll: workplace hazards of local government firefighters, 2009. Monthly Labor Review, 135, 18-25.
- [Background] Page, P., Frank, C.C., & Lardner, R. (2010). Assessment and Treatment of Muscle Imbalance: The Janda Approach. Champaign, IL: Human Kinetics.
- [Background] Peate WF, Bates G, Lunda K, Francis S, Bellamy K. Core strength: a new model for injury prediction and prevention. J Occup Med Toxicol. 2007 Apr 11;2:3. doi: 10.1186/1745-6673-2-3. PMID 17428333
- [Background] Perry FT, Koehle MS. Normative data for the functional movement screen in middle-aged adults. J Strength Cond Res. 2013 Feb;27(2):458-62. doi: 10.1519/JSC.0b013e3182576fa6. PMID 22561971
- [Background] Reiman, M.P., & Manske, R.C. (2009). Functional Testing in Human Performance. Champaign, IL: Human Kinetics.
- [Background] Seabury SA, McLaren CF. The Frequency, Severity, and Economic Consequences of Musculoskeletal Injuries to Firefighters in California. Rand Health Q. 2012 Sep 1;2(3):4. eCollection 2012 Fall. PMID 28083263
- [Background] TriData Corporation (2005). The Economic Consequences of Firefighter Injuries and their Prevention. Final Report. Arlington, VA: National Institute of Standards and Technology, U.S. Department of Commerce.